CLINICAL TRIAL: NCT01007942
Title: A Randomized Phase III, Double-blind, Placebo-controlled Multicenter Trial of Daily Everolimus in Combination With Trastuzumab and Vinorelbine, in Pretreated Women With HER2/Neu Over-expressing Locally Advanced or Metastatic Breast Cancer.
Brief Title: Daily Everolimus in Combination With Trastuzumab and Vinorelbine in HER2/Neu Positive Women With Locally Advanced or Metastatic Breast Cancer
Acronym: BOLERO-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRAD001W2301; 2008-008697-31 (EudraCT Number)
Record Dates: First submitted 2009-11-02; First posted 2009-11-04 (Estimated); Results first posted 2017-04-05 (Actual); Last update posted 2017-04-05 (Actual); Status verified 2017-02

CONDITIONS: HER2/Neu Over-expressing Locally Advanced Breast Cancer; Metastatic Breast Cancer
Keywords: Metastatic breast cancer; locally advanced breast cancer; HER2/neu positive breast cancer; HER2/neu over-expressing; progressive-free survival (PFS); over survival (OS); bolero; bolero 3; Breast cancer; everolimus; HER+; vinorelbine; herceptin; trastuzumab; RAD001
MeSH Terms: conditions — Breast Neoplasms | interventions — Everolimus; Vinorelbine; Trastuzumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Everolimus + vinorelbine + trastuzumab (Experimental): Oral everolimus (5 mg/day) + intravenous vinorelbine (25 mg/m2 weekly) + intravenous trastuzumab (2 mg/kg weekly following a 4 mg/kg loading dose on Day 1 of Cycle 1 only)
  Interventions: Drug: everolimus; Drug: vinorelbine; Drug: trastuzumab
- placebo + vinorelbine + trastuzumab (Placebo Comparator): Oral daily matching placebo + intravenous vinorelbine (25 mg/m2 weekly) + intravenous trastuzumab (2 mg/kg weekly following a 4 mg/kg loading dose on Day 1 of Cycle 1 only
  Interventions: Drug: Placebo; Drug: vinorelbine; Drug: trastuzumab

INTERVENTIONS:
Drug: everolimus — Oral everolimus was taken once 5 mg/day (2 × 2.5 mg tablets) and were packaged into blister packs.
  Other Names: RAD001
  Arms: Everolimus + vinorelbine + trastuzumab
Drug: Placebo — Oral everolimus placebo was taken once 5 mg/day (2 × 2.5 mg tablets) and were packaged into blister packs.
  Arms: placebo + vinorelbine + trastuzumab
Drug: vinorelbine — intravenous vinorelbine (25 mg/m2 weekly)
Drug: trastuzumab — intravenous trastuzumab (2 mg/kg weekly following a 4 mg/kg loading dose on Day 1 of Cycle 1 only)

SUMMARY:
This phase III, double-blind, placebo-controlled multinational study will assess the combination everolimus, vinorelbine, and trastuzumab compared to the combination vinorelbine and trastuzumab with respect to progressive-free survival and over survival in HER2/neu positive women with locally advanced or metastatic breast cancer who are resistant to trastuzumab and have been pre-treated with a taxane.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed invasive breast carcinoma with locally recurrent or radiological evidence of metastatic disease. Locally recurrent disease must not be amenable to resection with curative intent.
* HER2+ status defined as IHC 3+ staining or in situ hybridization positive
* Patients with resistance to trastuzumab
* Prior taxane therapy
* Patients with an ECOG performance status of 0 - 2
* Patients with measurable disease as per RECIST criteria
* Documentation of negative pregnancy test for patients of child bearing potential prior to enrollment within 7 days prior to randomization. Sexually active pre-menopausal women must use adequate contraceptive measures, excluding estrogen containing contraceptives, while on study;
* Patients must meet laboratory criteria defined in the study within 21 days prior to randomization

Exclusion Criteria:

* Prior mTOR inhibitors or vinca alkaloid agents for the treatment of cancer
* More than three prior chemotherapy lines for advanced disease.
* Symptomatic CNS metastases or evidence of leptomeningeal disease. Previously treated asymptomatic CNS metastases are allowed provided that the last treatment for CNS metastases was completed >8 weeks prior to randomization
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral everolimus
* Peripheral neuropathy ≥ grade 2 at randomization
* Active cardiac disease
* History of cardiac dysfunction
* Any malignancy within 5 years prior to randomization, with the exception of adequately treated in-situ carcinoma of the cervix uteri, basal or squamous cell carcinoma or non-melanomatous skin cancer
* Known hypersensitivity to any study medication
* Breastfeeding or pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 569 (Actual)
Dates: Start 2009-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (150):
- United States (43):
  - University of Arizona / Cancer Center AZ Onc Assoc, Tucson, Arizona
  - University of Arizona / Cancer Center Deptof Uof A/Arizona Cancer(3), Tucson, Arizona
  - University of California San Diego - Moores Cancer Center La Jolla - UCSD Moores Cancer, La Jolla, California
  - Rocky Mountain Cancer Centers RMCC, Greenwood Village, Colorado
  - Georgetown University/Lombardi Cancer Center Dept.of Lombardi CancerCtr (3), Washington D.C., District of Columbia
  - Comprehensive Cancer Center - Boca Raton Deerfield Beach, Boca Raton, Florida
  - Comprehensive Cancer Center - Boca Raton Dept.of BocaRatonCompCanCtr, Boca Raton, Florida
  - Florida Cancer Specialists DeptofFloridaCancerSpecialists, Fort Myers, Florida
  - Memorial Hospital Memorial Cancer Institute, Hollywood, Florida
  - MD Anderson Cancer Center - Orlando Dept.ofMDACC-Orlando(2), Orlando, Florida
  - Emory University School of Medicine/Winship Cancer Institute Dept.of WinshipCancerInst. (2), Atlanta, Georgia
  - North Shore University Health System NSU, Evanston, Illinois
  - Kansas City Cancer Center KCCC- South (2), Overland Park, Kansas
  - Maryland Oncology Hematology, Owning Mills, Maryland
  - Park Nicollet Institute Dept. of Park Nicollet, Saint Louis Park, Minnesota
  - St. Louis University Cancer Center SLU Cancer Center, St Louis, Missouri
  - University of Nebraska Medical Center Unv Nebraska Med Ctr (2), Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada CCC of Nevada Henderson (4), Las Vegas, Nevada
  - Nevada Cancer Institute Dept. of Nevada Cancer (3), Las Vegas, Nevada
  - Overlook Hospital - Carol G Simon Cancer Center Carol G Simon, Summit, New Jersey
  - Clinical Research Alliance Dept.ofArenaOncologyAssoc(2), Lake Success, New York
  - Duke University Medical Center Dept. of DUMC (2), Durham, North Carolina
  - Northwest Cancer Specialists Tutlatin, Portland, Oregon
  - University of Pittsburgh Cancer Institute DeptofMageeWomen'sHospital(2), Pittsburgh, Pennsylvania
  - The Jones Clinic Dept .of The Jones Clinic (3), Germantown, Tennessee
  - Sarah Cannon Research Institute Dept.ofSarahCannonCancerCtr(6), Nashville, Tennessee
  - Texas Cancer Center ( Medical City Dallas Hospital) Dept. of Texas Cancer Ctr. (2), Dallas, Texas
  - Texas Oncology Presbyterian Hospital (2), Dallas, Texas
  - Texas Oncology Texas Onc - Amarillo, Dallas, Texas
  - Texas Oncology Texas Oncology - Sammons, Dallas, Texas
  - Texas Oncology Midtown, Dallas, Texas
  - University of Texas Southwestern Medical Center University of TX SW Med Ctr(2), Dallas, Texas
  - University of Texas/MD Anderson Cancer Center SC-5, Houston, Texas
  - Baylor College of Medicine Baylor, Houston, Texas
  - Longview Cancer Center Longview Cancer Center (2), Longview, Texas
  - Cancer Care Centers of South Texas / HOAST CCC of So. TX- San Antonio(2), San Antonio, Texas
  - South Texas Oncology and Hematology, PA South Texas Oncology (2), San Antonio, Texas
  - Tyler Cancer Center Dept.ofTylerCancerCtr. (2), Tyler, Texas
  - Utah Cancer Specialists Utah Cancer (2), Salt Lake City, Utah
  - Virginia Cancer Specialists Fairfax No.VA (2), Fairfax, Virginia
  - Virginia Oncology Associates Dept. of VOA (2), Norfolk, Virginia
  - Swedish Cancer Institute Swedish Cancer Institute, Seattle, Washington
  - Green Bay Oncology Green Bay Oncology, Green Bay, Wisconsin
- Argentina (9):
  - Novartis Investigative Site, C A B A, Buenos Aires
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, Mar del Plata, Buenos Aires
  - Novartis Investigative Site, Quilmes, Buenos Aires
  - Novartis Investigative Site, Córdoba, Córdoba Province
  - Novartis Investigative Site, Posadas, Misiones Province
  - Novartis Investigative Site, Rosario, Sante Fe
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
  - Novartis Investigative Site, Rio Negro, Viedma
- Australia (6):
  - Novartis Investigative Site, Kogarah, New South Wales
  - Novartis Investigative Site, St Leonards, New South Wales
  - Novartis Investigative Site, South Brisbane, Queensland
  - Novartis Investigative Site, Southport, Queensland
  - Novartis Investigative Site, Hobart, Tasmania
  - Novartis Investigative Site, East Bentleigh, Victoria
- Belgium (4):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Namur
  - Novartis Investigative Site, Sint-Niklaas
- China (5):
  - Novartis Investigative Site, Shanghai, Shanghai Municipality
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Shanghai
- Czechia (3):
  - Novartis Investigative Site, Nový Jičín
  - Novartis Investigative Site, Olomouc
  - Novartis Investigative Site, Prague
- France (8):
  - Novartis Investigative Site, Bayonne
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Hyères
  - Novartis Investigative Site, La Chaussée-Saint-Victor
  - Novartis Investigative Site, La Roche-sur-Yon
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Saint-Brieuc Cédex
  - Novartis Investigative Site, Villejuif
- Germany (13):
  - Novartis Investigative Site, Mainz, Germany
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Gerlingen
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Homburg
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Minden
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Recklinghausen
  - Novartis Investigative Site, Velbert
- Greece (5):
  - Novartis Investigative Site, Athens, Greece
  - Novartis Investigative Site, Heraklion Crete, Greece
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Patra - RIO, GR
  - Novartis Investigative Site, Thessaloniki, GR
- Hungary (3):
  - Novartis Investigative Site, Győr, Hungary
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
- Israel (4):
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Italy (4):
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Sondrio, SO
- Japan (12):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Maebashi, Gunma
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kumamoto, Kumamoto
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Koto, Tokyo
- Mexico (2):
  - Novartis Investigative Site, León, Guanajuato
  - Novartis Investigative Site, Mexico City, Mexico City
- Poland (2):
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Warsaw
- Novartis Investigative Site, Singapore, Singapore, Singapore
- Slovakia (2):
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Košice
- Spain (12):
  - Novartis Investigative Site, Córdoba, Andalusia
  - Novartis Investigative Site, Jaén, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Barcelona, Barcelona
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Madrid, Madrid
  - Novartis Investigative Site, Majadahonda, Madrid
  - Novartis Investigative Site, San Cristóbal de La Laguna, Santa Cruz de Tenerife
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Zaragoza, Zaragoza
- Thailand (2):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Songkhla
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Ankara, Turkey
  - Novartis Investigative Site, Izmir, Turkey
  - Novartis Investigative Site, Fatih / Istanbul
- United Kingdom (7):
  - Novartis Investigative Site, Truro, Cornwall
  - Novartis Investigative Site, Surrey, England
  - Novartis Investigative Site, Bournemouth
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Plymouth

REFERENCES:
- [Derived] Andre F, O'Regan R, Ozguroglu M, Toi M, Xu B, Jerusalem G, Masuda N, Wilks S, Arena F, Isaacs C, Yap YS, Papai Z, Lang I, Armstrong A, Lerzo G, White M, Shen K, Litton J, Chen D, Zhang Y, Ali S, Taran T, Gianni L. Everolimus for women with trastuzumab-resistant, HER2-positive, advanced breast cancer (BOLERO-3): a randomised, double-blind, placebo-controlled phase 3 trial. Lancet Oncol. 2014 May;15(6):580-91. doi: 10.1016/S1470-2045(14)70138-X. Epub 2014 Apr 14. PMID 24742739

RESULTS

PARTICIPANT FLOW:
Recruitment Details: DCO ( Data cut-off) for patient disposition is 1-Apr-2015. Each Cycle = 21 days
Pre-assignment Details: 284 patients randomized to the Everolimus + trastuzumab + vinorelbine arm, 280 took drug. 285 patients randomized to the placebo + trastuzumab + vinorelbine arm, 282 too drug. A total of 569 were comprised to randomized total and 562 to safety.
Groups:
- Placebo + Vinorelbine + Trastuzumab: Oral daily matching placebo + intravenous vinorelbine (25 mg/m2 weekly) + intravenous trastuzumab (2 mg/kg weekly following a 4 mg/kg loading dose on Day 1 of Cycle 1 only)
Period: Overall Study
Arm/Group | Everolimus + Vinorelbine + Trastuzumab | Placebo + Vinorelbine + Trastuzumab
Started | 284 | 285
Completed | 3 (Pts completed= on treatment at time of DCO. Not Completed = ended treatment as per protocol.) | 7 (Pts completed= on treatment at time of DCO. Not Completed = ended treatment as per protocol.)
Not Completed | 281 | 278
Not completed — Adverse Event | 29 | 14
Not completed — Abnormal test procedure | 0 | 1
Not completed — Disease progression | 217 | 242
Not completed — New cancer therapy | 5 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 19 | 14
Not completed — Lost to Follow-up | 1 | 0
Not completed — Administrative problems | 2 | 0
Not completed — Death | 3 | 2
Not completed — Patients untreated | 4 | 3

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) consisted of all randomized patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Everolimus + Vinorelbine + Trastuzumab | Placebo + Vinorelbine + Trastuzumab | Total
Number analyzed (Participants) | 284 | 285 | 569
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (10.98) | 53.4 (11.00) | 53.8 (10.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 284 | 285 | 569
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progressive-free Survival (PFS) Per Investigator Assessment
Description: PFS was defined as the time from the date of randomization to the date of first radiologically documented tumor progression or death from any cause, whichever occurs first. PFS primary analysis performed when 415 events were reached. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Every 6 weeks until disease progression or death which ever occurred first up to about 41 months
Population: The Full Analysis Set (FAS) consisted of all randomized patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus + Vinorelbine + Trastuzumab | Placebo + Vinorelbine + Trastuzumab
Number analyzed (Participants) | 284 | 285
months | 7.00 [6.74 to 8.18] | 5.78 [5.49 to 6.90]
Statistical Analysis 1: Comparison: Everolimus + Vinorelbine + Trastuzumab vs Placebo + Vinorelbine + Trastuzumab; Test type: Superiority or Other; p = 0.0067, Log Rank; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.65 to 0.95]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from date of randomization to the date of death from any cause. Final OS was conducted when 388 deaths occurred.
Time Frame: Every 3 months until death up to 41 months
Population: The Full Analysis Set (FAS) consisted of all randomized patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus + Vinorelbine + Trastuzumab | Placebo + Vinorelbine + Trastuzumab
Number analyzed (Participants) | 284 | 285
months | 23.46 [20.01 to 28.81] | 24.08 [21.49 to 27.63]

3. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants whose best overall response was either complete response (CR) or partial response (PR) according to RECIST version 1.0. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Every 6 weeks until disease progression or death which ever occurred first up to about 41 months
Population: The Full Analysis Set (FAS) consisted of all randomized patients.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Everolimus + Vinorelbine + Trastuzumab | Placebo + Vinorelbine + Trastuzumab
Number analyzed (Participants) | 284 | 285
Percentage of participants | 40.8 [35.1 to 46.8] | 37.2 [31.6 to 43.1]

4. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR was defined as the percentage of participants whose best overall response, according to RECIST, was either complete response (CR), a partial response (PR) or stable disease (SD) lasting for at least 24 weeks. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; SD = Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for PD; PD = At least a 20% increase in the sum of the longest diameter of all measured target lesions, taking as reference the smallest sum of longest diameter of all target lesions recorded at or after baseline.
Time Frame: Every 6 weeks until disease progression or death which ever occurred first up to about 41 months
Population: The Full Analysis Set (FAS) consisted of all randomized patients.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Everolimus + Vinorelbine + Trastuzumab | Placebo + Vinorelbine + Trastuzumab
Number analyzed (Participants) | 284 | 285
Percentage of participants | 59.2 [53.2 to 64.9] | 53.3 [47.4 to 59.2]

5. Secondary Outcome: Median Time to Deterioration of the ECOG Performance Status Score
Description: Time to deterioration of ECOG performance status score was summarized at time of assessment. ECOG (Eastern Cooperative Oncology Group)performance scale is a standard criteria for measuring how treatment of cancer impacts their level of functioning in terms of their ability to care for themselves, daily activity, & physical ability (walking, working, etc.). Scale score ranges from 0 to 5, 5 being the worst. ECOG scale index: 0 - Fully active, able to carry on all pre-disease performance without restriction. 1 - Restricted in physically strenuous activity but ambulatory & able to carry out work of a light or sedentary nature, e.g., light housework, office work. 2 - Ambulatory & capable of all self-care but unable to carry out any work activities. Up & about more than 50% of waking hours. 3 - Capable of only limited self-care, confined to bed or chair more than 50% of waking hours. 4 - Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair. 5 - Dead
Time Frame: baseline, until disease progression or death up to about 41 months
Population: The Full Analysis Set (FAS) consisted of all randomized patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus + Vinorelbine + Trastuzumab | Placebo + Vinorelbine + Trastuzumab
Number analyzed (Participants) | 284 | 285
months | 32.66 [17.68 to 32.66] | 21.55 [12.48 to NA] — N/A = data could not be analyzed at later time points due to the low number of patients.

6. Secondary Outcome: PRO: Time to Deterioration in Global Health Status/QoL Domain Score of the European Organization for the Research and Treatment of Cancer (EORTC)-Core Quality of Life Questionnaire (QLQ-C30) (by at Least 10%)
Description: PRO = patient reported outcomes; Time to deterioration (≥ 10% worsening from baseline), in the global health status of EORTC QLQ-C30 scale was done in the 3 functional scales (emotional, physical, & social functioning [EF, PF, & SF]). It contains 30 items & is composed of multi-item scales & single-item measures. These include 5 functional scales (physical, role, emotional, social & cognitive functioning), 3 symptom scales (fatigue, pain, nausea, & vomiting), a global health status/QoL scale, and 6 single items (dyspnea, diarrhea, constipation, anorexia, insomnia & financial impact). Each of the multi-item scale includes a different set of items - no item occurs in more than 1 scale. Each item in the EORTC QLQ-C30 has 4 response categories (1=Not at all, 2= A little, 3= Quite a bit, 4= Very much) with the higher number representing a worse outcome. The global health domain score of the QLQ-C30 questionnaire was pre-specified as the primary QoL domain of interest & disclosed here.
Time Frame: Baseline, until disease progression or death up to about 41 months
Population: The Full Analysis Set (FAS) consisted of all randomized patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus + Vinorelbine + Trastuzumab | Placebo + Vinorelbine + Trastuzumab
Number analyzed (Participants) | 284 | 285
months
  Deterioration - global QoL domain by at least 10% | 8.31 [6.93 to 11.53] | 7.29 [5.55 to 10.38]
  Deterioration in the PF domain by at least 10% | 11.96 [8.31 to 14.09] | 12.48 [8.31 to 20.86]
  Deterioration in the EF domain by at least 10% | 15.18 [9.20 to 17.28] | 12.45 [9.69 to 16.36]
  Deterioration in the SF domain by at least 10% | 11.33 [8.18 to 14.52] | 13.11 [8.31 to 19.32]

7. Secondary Outcome: Everolimus Blood Concentrations by Leading Dose and Time Point
Description: Pre-dose (Cmin) and 2 hours post-dose (C2h) everolimus PK blood samples were collected at Cycle 2 Day 1. Only valid everolimus PK blood samples collected at steady state were used in the analyses.
Time Frame: Cycle 2, Day 1
Population: The Safety Set consisted of all patients who received at least one dose of the study treatment and who had at least one valid post-baseline safety assessment.
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Everolimus 2.5 mg: Oral everolimus of 2.5 mg/day
- Everolimus: Oral everolimus of 5 mg/day
Arm/Group | Everolimus 2.5 mg | Everolimus
Number analyzed (Participants) | 10 | 43
ng/ml
  Pre-dose (Cmin) (n: 7, 32) | 2.928 (2.6197) | 5.652 (4.1006)
  2 hours post administration (C2h) (n:10, 43) | 13.035 (6.6842) | 22.005 (13.3800)

8. Secondary Outcome: Vinorelbine Blood Concentrations by Leading Dose and Time Point
Description: Pre-infusion (Cmin) and end of infusion (C2h) vinorelbine PK blood samples were collected at Cycle 2 Day 1. Only valid vinorelbine PK blood samples collected at steady state were used in the analyses.
Time Frame: Cycle 2, Day 1
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Everolimus Placebo: Oral placebo everolimus of 5 mg/day
Arm/Group | Everolimus | Everolimus Placebo
Number analyzed (Participants) | 76 | 64
ng/ml
  Pre-infusion - dose (Cmin) (n: 76, 64) | 11.085 (66.8551) | 0.061 (0.4888)
  End of infusion (Cmax) (n: 58, 49) | 867.147 (971.3057) | 1068.51 (1145.860)

9. Secondary Outcome: Trastuzumab Blood Concentrations by Leading Dose and Time Point
Description: Pre-infusion (Cmin) and end of infusion (C2h) trastuzumab PK blood samples were collected at Cycle 3 Day 1. Only valid trastuzumab PK blood samples collected at steady state were used in the analyses.
Time Frame: Cycle 3, Day 1
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Everolimus | Everolimus Placebo
Number analyzed (Participants) | 74 | 59
ng/ml
  Pre-infusion - dose (Cmin) (n: 73, 57) | 23.351 (6.3344) | 24.526 (7.9960)
  End of infusion (Cmax) (n: 75, 59) | 64.279 (27.8549) | 60.576 (15.5198)

ADVERSE EVENTS:
Groups:
- Everolimus + Trastuzumab + Vinorelbine: Oral everolimus (5 mg/day) + intravenous vinorelbine (25 mg/m2 weekly) + intravenous trastuzumab (2 mg/kg weekly following a 4 mg/kg loading dose on Day 1 of Cycle 1 only)
- Placebo + Trastuzumab + Vinorelbine: Oral daily matching placebo + intravenous vinorelbine (25 mg/m2 weekly) + intravenous trastuzumab (2 mg/kg weekly following a 4 mg/kg loading dose on Day 1 of Cycle 1 only)
Arm/Group | Everolimus + Trastuzumab + Vinorelbine | Placebo + Trastuzumab + Vinorelbine
Serious Adverse Events (participants affected / at risk) | 122/280 | 58/282
Other Adverse Events (participants affected / at risk) | 280/280 | 280/282
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus + Trastuzumab + Vinorelbine (N=280) | Placebo + Trastuzumab + Vinorelbine (N=282)
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 10 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 30 | 4
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 3 | 0
Neutropenia (Blood and lymphatic system disorders) | 12 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cataract (Eye disorders) | 2 | 1
Cataract subcapsular (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastric perforation (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 2 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 1
Neutropenic colitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 9 | 1
Vomiting (Gastrointestinal disorders) | 5 | 2
Asthenia (General disorders) | 0 | 1
Chills (General disorders) | 2 | 0
Device dislocation (General disorders) | 0 | 1
Extravasation (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 3 | 2
Hyperpyrexia (General disorders) | 0 | 1
Hyperthermia (General disorders) | 0 | 1
Inflammation (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 2 | 0
Pyrexia (General disorders) | 13 | 5
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Hepatic mass (Hepatobiliary disorders) | 0 | 1
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0
Abscess jaw (Infections and infestations) | 0 | 1
Aspergillus infection (Infections and infestations) | 1 | 0
Bronchiolitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 4 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 3 | 1
Device related sepsis (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Furuncle (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0
Gastroenteritis clostridial (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 2 | 0
Klebsiella bacteraemia (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 2 | 0
Neutropenic infection (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 2 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Peritonsillar abscess (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 2 | 0
Pneumocystis jirovecii infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 8 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 3 | 0
Sinusitis (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 2
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain oedema (Nervous system disorders) | 1 | 1
Disturbance in attention (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 3
Hydrocephalus (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0
Neurological symptom (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 3 | 1
Somnolence (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 3 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 2
Shock (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus + Trastuzumab + Vinorelbine (N=280) | Placebo + Trastuzumab + Vinorelbine (N=282)
Anaemia (Blood and lymphatic system disorders) | 137 | 85
Febrile neutropenia (Blood and lymphatic system disorders) | 17 | 7
Leukopenia (Blood and lymphatic system disorders) | 126 | 105
Neutropenia (Blood and lymphatic system disorders) | 226 | 196
Thrombocytopenia (Blood and lymphatic system disorders) | 39 | 6
Abdominal pain (Gastrointestinal disorders) | 45 | 52
Abdominal pain upper (Gastrointestinal disorders) | 34 | 40
Constipation (Gastrointestinal disorders) | 84 | 88
Diarrhoea (Gastrointestinal disorders) | 108 | 88
Dry mouth (Gastrointestinal disorders) | 14 | 7
Dyspepsia (Gastrointestinal disorders) | 21 | 25
Mouth ulceration (Gastrointestinal disorders) | 32 | 6
Nausea (Gastrointestinal disorders) | 98 | 105
Stomatitis (Gastrointestinal disorders) | 174 | 78
Vomiting (Gastrointestinal disorders) | 57 | 59
Asthenia (General disorders) | 74 | 57
Chills (General disorders) | 18 | 18
Fatigue (General disorders) | 124 | 119
Non-cardiac chest pain (General disorders) | 11 | 20
Oedema peripheral (General disorders) | 39 | 23
Pain (General disorders) | 20 | 20
Pyrexia (General disorders) | 107 | 65
Nasopharyngitis (Infections and infestations) | 37 | 29
Upper respiratory tract infection (Infections and infestations) | 38 | 26
Urinary tract infection (Infections and infestations) | 26 | 18
Alanine aminotransferase increased (Investigations) | 37 | 26
Aspartate aminotransferase increased (Investigations) | 33 | 22
Ejection fraction decreased (Investigations) | 17 | 5
Gamma-glutamyltransferase increased (Investigations) | 29 | 23
Haemoglobin decreased (Investigations) | 22 | 18
Neutrophil count decreased (Investigations) | 14 | 8
Weight decreased (Investigations) | 83 | 47
White blood cell count decreased (Investigations) | 17 | 23
Decreased appetite (Metabolism and nutrition disorders) | 94 | 49
Hypercholesterolaemia (Metabolism and nutrition disorders) | 26 | 12
Hyperglycaemia (Metabolism and nutrition disorders) | 26 | 15
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 23 | 9
Hypokalaemia (Metabolism and nutrition disorders) | 34 | 19
Arthralgia (Musculoskeletal and connective tissue disorders) | 48 | 36
Back pain (Musculoskeletal and connective tissue disorders) | 37 | 46
Bone pain (Musculoskeletal and connective tissue disorders) | 28 | 24
Muscle spasms (Musculoskeletal and connective tissue disorders) | 31 | 47
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 16 | 12
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 14 | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 39 | 31
Pain in extremity (Musculoskeletal and connective tissue disorders) | 42 | 44
Dizziness (Nervous system disorders) | 31 | 24
Dysgeusia (Nervous system disorders) | 32 | 17
Headache (Nervous system disorders) | 74 | 62
Hypoaesthesia (Nervous system disorders) | 15 | 7
Neuropathy peripheral (Nervous system disorders) | 27 | 41
Paraesthesia (Nervous system disorders) | 21 | 21
Peripheral sensory neuropathy (Nervous system disorders) | 25 | 17
Anxiety (Psychiatric disorders) | 13 | 18
Insomnia (Psychiatric disorders) | 34 | 27
Cough (Respiratory, thoracic and mediastinal disorders) | 84 | 55
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 51 | 40
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 64 | 38
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 27 | 27
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 17 | 9
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 17 | 14
Alopecia (Skin and subcutaneous tissue disorders) | 22 | 29
Pruritus (Skin and subcutaneous tissue disorders) | 16 | 29
Rash (Skin and subcutaneous tissue disorders) | 71 | 54
Hot flush (Vascular disorders) | 4 | 16
Hypertension (Vascular disorders) | 24 | 10
Phlebitis (Vascular disorders) | 14 | 18

LIMITATIONS AND CAVEATS:
All randomized patients were included in the FAS. Seven patients (4 in the everolimus arm & 3 in the placebo arm) were randomized but never received treatment & were therefore excluded from the Safety Set.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.